CLINICAL TRIAL: NCT01701362
Title: A Randomized Double Blind Placebo Controlled Parallel Group Study Of The Efficacy And Safety Of Pregabalin (Bid) In Subjects With Post-traumatic Peripheral Neuropathic Pain
Brief Title: Placebo-controlled Safety and Efficacy Study of Pregabalin in Subjects With Post-traumatic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081279; 2012-003304-12 (EudraCT Number)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2017-04

CONDITIONS: Neuropathic Pain
Keywords: post-traumatic peripheral neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin (Active Comparator)
  Interventions: Drug: pregabalin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — capsules, 150-600 mg/day administered in divided doses twice a day for 15 weeks after randomization
  Other Names: Lyrica, PD-144723
  Arms: pregabalin
Drug: placebo — capsules, placebo for pregabalin administered in divided doses twice a day for 15 weeks after randomization
  Arms: placebo

SUMMARY:
This study is designed to investigate if pregabalin is effective in treating neuropathic (nerve) pain resulting from peripheral nerve trauma due to a traumatic or surgical event such as, for example, motor vehicle accident, fall, sports injury, knee or hip replacement, hernia repair, thoracotomy, mastectomy, focal/localized burns or crush injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have chronic peripheral neuropathic pain present for than 6 months after a traumatic or surgical event such as, for example, motor vehicle accident, fall, sports injury, knee or hip replacement, hernia repair, thoracotomy, mastectomy, focal/localized burns or crush injury.
* Subjects must be literate and have the ability (unaided) to understand and use the interactive voice response system (IVRS), have daily access to a telephone in order to complete the IVRS assessments each day, perform telephone visits and complete all required assessments/forms.
* Subjects must have sufficient post-traumatic neuropathic pain at screening and baseline.

Exclusion Criteria:

* Subjects with neuropathic pain due to diabetic peripheral neuropathy (DPN), post herpetic neuralgia (PHN), HIV, trigeminal neuralgia (TGN), carpal tunnel syndrome (CTS) or with central neuropathic pain (for example, due to spinal cord injury) or with Complex Regional Pain Syndrome (CRPS, Type I or Type II).
* Subjects with other pain that may confound assessment or self-evaluation of the peripheral neuropathic pain.
* Subjects who have failed pregabalin treatment due to lack of efficacy with an adequate course of therapy at doses greater than or equal to 150 mg/day, who have previously participated in a pregabalin clinical trial or who have been treated with pregabalin at any time during the 6 month period prior to screening.
* Subjects with epilepsy; pernicious anemia; hematological illnesses; known HIV infection; any clinically unstable cardiovascular (including a myocardial infarction [heart attack] in the 3 months prior to screening), hematological, autoimmune, endocrine, renal, hepatic (including chronic hepatitis B, hepatitis B within the 3 months prior to screening) respiratory, or gastrointestinal disease; symptomatic peripheral vascular disease including intermittent claudication; uncontrolled diabetes mellitus; untreated hypothyroidism.
* Subjects with a diagnosis of DSM-IV TR Axis I disorder (including, for example, schizophrenia, bipolar disorder) with the exceptions of Generalized Anxiety Disorder (GAD) or major depression that is clinically stable.
* Subjects considered at risk of suicide or self-harm based on investigator judgment and/or details of a risk assessment.
* Use of prohibited medications in the absence of appropriate washout periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (155):
- United States (104):
  - Tennesse Valley Pain Consultants, Huntsville, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Neuromuscular Research Center, Phoenix, Arizona
  - Quality of Life Medical & Research Centers, LLC, Tucson, Arizona
  - Advanced Rx Clinical Research, Artesia, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - NervePro Medical Corp., Irvine, California
  - University of California, Irvine, Irvine, California
  - Clinical and Translational Research Institute, La Jolla, California
  - Alliance Research Centers, Laguna Hills, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Center For United Research, Inc., Lakewood, California
  - University of Southern California, Los Angeles, California
  - USC I.D.S. Pharmacy, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - North County Clinical Research, Oceanside, California
  - Allied Clinical Research, Roseville, California
  - Northern California Research, Sacramento, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Colorado Clinic, Boulder, Colorado
  - Mountain View Clinical Research Inc., Denver, Colorado
  - St. Luke's Medical Clinic, Fort Collins, Colorado
  - Investigational Drug Services, The George Washington University Medical Center, Washington D.C., District of Columbia
  - The George Washington University Medical Center (Department of Neurology), Washington D.C., District of Columbia
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Advance Medical Research, Clearwater, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - Aga Clinical Trials, Hialeah, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - Research in Miami, Inc., Hialeah, Florida
  - Homestead Medical Research , Inc., Homestead, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Compass Research, LLC, Orlando, Florida
  - A-One Family Practice, Ormond Beach, Florida
  - Aba Family Medicine, LLC, Ormond Beach, Florida
  - Ribo Research, LLC dba Peninsula Resarch, Ormond Beach, Florida
  - Comprehensive Pain Care of South Florida, Royal Palm Beach, Florida
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - Meridien Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Advanced Internal Medicine, PC, Stockbridge, Georgia
  - Research 1 Clinical Research Network, Inc. (Administrative Office Only), Stockbridge, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Chicago Anesthesia Associates, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, Overland Park, Kansas
  - Otri-Med Corporation, Edgewood, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Centex Studies, Inc, Lake Charles, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - University of Rochester, Translational Pain Research, Rochester, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Northern Ohio Neurosciences, LLC, Bellevue, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Northwest Ohio Research Center, LLC, Toledo, Ohio
  - Robert L Kalb, M.D, Inc, Toledo, Ohio
  - Cor Clinical Research, Llc, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network, Inc., Portland, Oregon
  - Allegheny Pain Management, P.C., Altoona, Pennsylvania
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Piedmont Comprehensive Pain Management Group, LLC, Greenville, South Carolina
  - Pharmacum Biomedical Research, Greenville, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Dallas Pain Consultants, Dallas, Texas
  - FutureSearch Trials of Dallas, L. P., Dallas, Texas
  - Abigail R. Neiman, MD, PA, Houston, Texas
  - Agadadash Kuliev, MD, PA, Houston, Texas
  - Biopharma Informatic Inc. Research Center, Houston, Texas
  - Medstar Clinical Research Associates, Houston, Texas
  - ClinRx Research, LLC, Richardson, Texas
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Sealy Urgent Care Center and Medical Clinic, Sealy, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc./Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewish Research, Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - Integrated Neurology Services , PLLC, Arlington, Virginia
  - IntegraTrials, LLC, Arlington, Virginia
  - Washington Center for Pain Management LLC, Bellevue, Washington
  - Northwest Clinical Research Center, Bellevue, Washington
  - Washington Center for Pain Management LLC, Edmonds, Washington
  - Washington Center for Pain Management LLC, Everett, Washington
  - Washington Center for Pain Management LLC, Renton, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
- Bulgaria (6):
  - MHAT Puls AD, Blagoevgrad
  - MHAT "Avis Medika", Pleven
  - MHAT "Sv.Pantaleymon", Pleven
  - DCC Akta Medika Ltd., Sevlievo
  - UMHAT Aleksandrovska, Sofia
  - DCC "Sveta Anna"EOOD, Sofia
- Canada (4):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - NRK Medical Research Clinic (Adminstrative Office Only), London, Ontario
  - NRK Medical Research Clinic, London, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
- General Hospital "dr. Ivo Pedisic", Sisak, Croatia
- Glostrup Hospital, Glostrup Municipality, Denmark
- Germany (12):
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Praxis für Spezielle Schmerztherapie und Palliativmedizin, Böhlen, Saxony
  - medamed GmbH Studienambulanz, Leipzig, Saxony
  - pro scientia med im MARE Klinikum, Kiel-Kronshagen, Schleswig-Holstein
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Synexus Clinical Research GmbH, Frankfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Gemeinschaftspraxis für Schmerz- und Psychotherapie, Hamburg
  - Synexus Clinical Research GmbH, Leipzig
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (3):
  - Synexus Magyarorszag Kft., Budapest
  - UNO Medical Trials Kft, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
- Poland (7):
  - Niepubliczny Zaklad Opieki Zdrowotnej "Przychodnia Morena" Sp. z.o.o., Gdansk
  - "SYNEXUS POLSKA" Sp. z o.o. Oddzial w Gdyni, Gdynia
  - "Synexus Polska" Sp. z o.o. Oddzial W Katowicach, Katowice
  - Malopolskie Centrum Medyczne S.C., Krakow
  - NZOZ IGNIS dr n. med. Alicja Lobinska, Świdnik
  - "SYNEXUS Polska" Sp. z o.o. ODDZIAL W WARSZAWIE, Warsaw
  - "SYNEXUS POLSKA" Sp. z o.o. Odzial we Wroclawiu, Wroclaw
- Ponce School of Medicine, CAIMED Center, Ponce, Puerto Rico
- Romania (6):
  - Centrul Medical Sana, Bucharest
  - Clubul Sanatatii SRL, Campulung Muscel
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Spitalul Clinic Municipal Dr. Gavril Curteanu Oradea,Sectia Neurologie I, Oradea
  - Spitalul Clinic Judetean de Urgenta Sibiu,Sectia Neurologie, Sibiu
  - Spitalul Clinic Judetean de Urgenta Targu-Mures , Sectia Neurologie II, Târgu Mureş
- South Africa (4):
  - Welkom Clinical Trial Centre, Welkom, Free State
  - Synexus SA - Stanza Clinical Research Centre, Pretoria, Gauteng
  - Synexus SA - Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Synexus SA - Roodepoort Medicross Clinical Research Centre, Roodeport, Gauteng
- Seoul National University Hospital, Seoul, South Korea
- Sweden (5):
  - Ladulaas Kliniken, Borås
  - CTC, Gothia Forum, Sahlgrenska Universitetssjukhus, Gothenburg
  - Probare, Lund
  - Pharmasite, Malmo
  - Bragee Medect AB, Stockholm

REFERENCES:
- [Derived] Markman J, Resnick M, Greenberg S, Katz N, Yang R, Scavone J, Whalen E, Gregorian G, Parsons B, Knapp L. Efficacy of pregabalin in post-traumatic peripheral neuropathic pain: a randomized, double-blind, placebo-controlled phase 3 trial. J Neurol. 2018 Dec;265(12):2815-2824. doi: 10.1007/s00415-018-9063-9. Epub 2018 Sep 21. PMID 30242745
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081279&StudyName=Placebo-controlled%20safety%20and%20efficacy%20study%20of%20pregabalin%20in%20subjects%20with%20post-traumatic%20peripheral%20neuropathic%20pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 187 centers participated in the study in 14 countries.
  During screening, with the exception of daily pain score data that was collected to determine participants eligibility, no participants were treated with active drug and no efficacy data were collected. Only safety and no efficacy data was collected during the taper period.
Pre-assignment Details: Participants had clinic visits at screening, randomization, and during the treatment period, and a phone contact for follow-up after the last taper dose. All the eligible participants were randomly assigned (1:1) to 15 weeks of treatment with Pregabalin or Placebo.
Groups:
- Pregabalin: Participants randomized to receive pregabalin: a 3-week dose optimization phase followed by 150 mg, 300 mg, 450 mg or 600 mg per day dosing 12-week maintenance phase.
- Placebo: Participants randomized to receive placebo
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 275 | 267
TREATED | 274 | 265
Completed | 233 | 211
Not Completed | 42 | 56
Not completed — Adverse events not related to study drug | 1 | 6
Not completed — Adverse events related to study drug | 12 | 10
Not completed — Protocol Violation | 5 | 3
Not completed — No longer willing to participate | 8 | 14
Not completed — Lost to Follow-up | 6 | 9
Not completed — Insufficient clinical response | 6 | 6
Not completed — Death | 0 | 1
Not completed — Randomized but not treated | 1 | 2
Not completed — Reasons other than those mentioned above | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 274 | 265 | 539
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (12.9) | 53.4 (12.7) | 53.1 (12.8)
Age, Customized [Number; unit: Participants]
  18 - 44 years | 59 | 61 | 120
  45 - 64 years | 163 | 154 | 317
  >=65 years | 52 | 50 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 134 | 266
  Male | 142 | 131 | 273

OUTCOME MEASURES:

1. Primary Outcome: Baseline Mean Pain Score
Description: This is based on the daily pain dairy and is defined as the baseline mean pain diary score. The Daily Pain Diary consists of an 11-point numeric rating scale (NRS) ranging from 0 ("no pain") to 10 ("worst possible pain"). Subjects describe their pain during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: Baseline
Population: Intent to Treat (ITT) population: all randomized participants who took at least one dose of study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
units on a scale | 6.41 (1.30) | 6.54 (1.30)

2. Primary Outcome: Change From Baseline to Week 15 in Weekly Mean Pain Score
Description: This is based on the daily pain diary and is defined as the change from baseline to week 15 in mean pain diary score. The Daily Pain Diary consists of an 11-point numeric rating scale (NRS) ranging from 0 ("no pain") to 10 ("worst possible pain"). Subjects describe their pain during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: up to Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
units on a scale | -2.12 (0.15) | -1.90 (0.16)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1823, Mixed Model Repeated Measures Analysis; Mixed Model Repeated Measures = MMRM; least squares mean difference = -0.22, 95% CI [-0.54 to 0.10], Standard Error of Mean 0.16 — MMRM analysis includes fixed categorical effects of treatment, country, trauma type, visit week, treatment-by-visit interaction, and fixed continuous effect of baseline value. Missing mean pain scores imputed by multiple imputation method

3. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 15
Description: A self administered instrument that measures changes in participants' overall status on a scale ranging from 1 (very much improved) to 7 (very much worse). The PGIC is based on the Clinical Global Impression of Change, which is a validated scale.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 258 | 246
Participants
  Very much improved | 52 | 41
  Much improved | 105 | 79
  Minimally improved | 61 | 62
  No change | 34 | 51
  Minimally worse | 5 | 9
  Much worse | 0 | 4
  Very much worse | 1 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — The p-value is derived from CMH test, stratified for pooled center and trauma type and excludes missing values

4. Secondary Outcome: Change From Baseline in Overall Weekly Mean Sleep Interference Score (SIRS)
Description: This is an 11-point NRS ranging from 0 ("pain does not interfere with sleep") to 10 ("pain completely interferes with sleep" [unable to sleep due to pain]). Participants describe how pain has interfered with their sleep during the past 24 hours. Please note that the data for Baseline (raw scores) have been included in the below table to read the change from Baseline data in context.
  Note: Weekly mean SIRS scores were derived from the daily sleep diary and calculated as the mean of the available scores in the 7 days. Generally, week 'n' mean SIRS scores were defined as the mean of the 7 daily diary SIRS scores from Day 2+7 (n-1) to Day 1+7*n. For participants with multiple diary scores collected on the same day, the average of all non-missing scores for that day was used in any analyses or data listings.
  "Overall" is the pooled average sleep interference score for each subject across all post-baseline/randomization weeks.
Time Frame: up to Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
units on a scale
  Baseline (raw scores) (N = 274, 265) | 4.97 (2.30) | 4.99 (2.27)
  Week 1 (N = 260, 258) | -0.66 (1.10) | -0.28 (0.91)
  Week 2 (N = 254, 244) | -1.15 (1.51) | -0.81 (1.27)
  Week 3 (N = 252, 245) | -1.55 (1.73) | -1.14 (1.45)
  Week 4 (N = 245, 229) | -1.73 (1.80) | -1.30 (1.63)
  Week 5 (N = 241, 226) | -1.87 (1.87) | -1.40 (1.68)
  Week 6 (N = 244, 227) | -1.94 (1.95) | -1.46 (1.79)
  Week 7 (N = 240, 216) | -2.01 (1.99) | -1.50 (1.78)
  Week 8 (N = 236, 212) | -2.05 (2.00) | -1.52 (1.76)
  Week 9 (N = 232, 214) | -2.09 (1.99) | -1.55 (1.86)
  Week 10 (N = 229, 212) | -2.04 (2.11) | -1.55 (1.83)
  Week 11 (N = 230, 211) | -2.09 (2.05) | -1.64 (1.79)
  Week 12 (N = 227, 209) | -2.17 (2.06) | -1.68 (1.89)
  Week 13 (N = 225, 204) | -2.19 (2.06) | -1.70 (1.90)
  Week 14 (N = 222, 208) | -2.19 (2.16) | -1.79 (1.89)
  Week 15 (N = 196, 186) | -2.13 (2.17) | -1.83 (1.87)
  Overall (N = 269, 262) | -1.83 (1.93) | -1.37 (1.71)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0119, Mixed Model Repeated Measures Analysis; Analyzed for treatment, center, trauma type, week & treatment-by-week interaction and fixed continuous effect of baseline value on the ITT population; least square mean difference = -0.35, 95% CI [-0.62 to -0.08], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; p = 0.0135, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.34, 95% CI [-0.62 to -0.07], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0028, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.42, 95% CI [-0.69 to -0.14], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0016, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.44, 95% CI [-0.72 to -0.17], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0007, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.48, 95% CI [-0.75 to -0.20], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; p = 0.0006, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.48, 95% CI [-0.76 to -0.21], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7; Test type: Superiority or Other; p = 0.0008, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.48, 95% CI [-0.75 to -0.20], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; p = 0.0003, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.52, 95% CI [-0.79 to -0.24], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 9; Test type: Superiority or Other; p = 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.54, 95% CI [-0.82 to -0.26], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Week 10; Test type: Superiority or Other; p = 0.0005, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.49, 95% CI [-0.77 to -0.22], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0007, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.48, 95% CI [-0.76 to -0.20], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.54, 95% CI [-0.82 to -0.27], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Week 13; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.56, 95% CI [-0.84 to -0.28], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Week 14; Test type: Superiority or Other; p = 0.0005, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.50, 95% CI [-0.78 to -0.22], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Week 15; Test type: Superiority or Other; p = 0.0031, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.43, 95% CI [-0.71 to -0.14], Standard Error of Mean 0.15
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Overall; Test type: Superiority or Other; p = 0.0001, Mixed Model Repeated Measures Analysis; [statistical method as in outcome 4, analysis 1]; least square mean difference = -0.47, 95% CI [-0.71 to -0.23], Standard Error of Mean 0.12

5. Secondary Outcome: Change From Baseline in Pain Severity Index (Brief Pain Inventory-short Form [BPI-sf])
Description: A self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24 hour period prior to evaluation. The BPI-sf consists of 5 questions. Four items measure pain on 11-point response scales from 0 (No Pain) to 10 (Pain as bad as you can imagine). In the above scale, score 0 indicates the better outcome whereas score 10 indicates the worse outcome.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 258 | 246
units on a scale | -2.40 (0.13) [-8.3 to 2.5] | -1.95 (0.13) [-6.5 to 2.5]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0050, ANCOVA; This secondary endpoint has been analyzed using ANCOVA with model terms of treatment, center, trauma type and baseline value on the ITT population; least squares mean difference = -0.46, 95% CI [-0.77 to -0.14], Standard Error of Mean 0.16

6. Secondary Outcome: Change From Baseline in Pain Interference Index (BPI-sf)
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24 hour period prior to evaluation.
  It consists of 7 sub-questions that evaluates the level of pain interference with daily functioning on 11-point response scales from 0 (does not interfere) to 10 (completely interferes).
  The BPI-sf pain interference index was calculated as average of the seven individual pain interference scores.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
units on a scale | -1.72 (0.13) [-1.97 to -1.46] | -1.33 (0.13) [-1.59 to -1.07]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0168, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI [-0.70 to -0.07], Standard Error of Mean 0.16

7. Secondary Outcome: Change From Baseline to Endpoint in Quality of Life Using EuroQol (EQ-5D) Health State Profile Scores
Description: A self-administered questionnaire designed to assess health related quality of life in terms of a single index value or utility score. There are 5 dimensions: mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression. Each dimension is rated on a 3 point response scale and the scores are combined to form a single index value between 0 and 1 with higher scores being more positive (better health status). The EQ-5D was completed by the subject at week-0 and week-15/ET where 30% responder and 50% responder status would be defined for each participants based on the percent change from baseline (week 0/Randomization) to each visit week in mean pain score and participant global impression of change (PGIC). PGIC is a self-administered instrument that measures change in participant's overall status on a scale ranging from 1 (very much improved) to 7 (very much worse). It is based on the Clinical Global Impression of Change CGIC), which is a validated scale.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Units on a scale
  Mobility | -0.10 (0.03) [-0.16 to -0.05] | -0.09 (0.03) [-0.15 to -0.03]
  Self-care | -0.08 (0.02) [-0.12 to 0.04] | -0.06 (0.02) [-0.11 to -0.02]
  Usual activities | -0.12 (0.03) [-0.19 to -0.05] | -0.13 (0.04) [-0.20 to -0.06]
  Pain/Discomfort | -0.35 (0.03) [-0.42 to -0.28] | -0.29 (0.04) [-0.36 to -0.22]
  Anxiety/Depression | 0.01 (0.03) [-0.05 to 0.07] | -0.02 (0.03) [-0.08 to 0.04]
  Dolan 1997 Index Score | 0.12 (0.01) | 0.11 (0.01)
  Dolan 2001 Index Score | -0.13 (0.02) | -0.12 (0.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; This statistical analysis is for mobility; Test type: Superiority or Other; p = 0.6841, ANCOVA; This sub-score has been analyzed using ANCOVA with model terms of treatment, center, trauma type and baseline value on the ITT population; least squares mean difference = -0.01, 95% CI [-0.09 to 0.06], Standard Error of Mean 0.037
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; This statistical analysis is for self-care; Test type: Superiority or Other; p = 0.6564, ANCOVA; [statistical method as in outcome 7, analysis 1]; least squares mean difference = -0.01, 95% CI [-0.07 to 0.04], Standard Error of Mean 0.029
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; This statistical analysis is for usual activities; Test type: Superiority or Other; p = 0.8590, ANCOVA; [statistical method as in outcome 7, analysis 1]; least squares mean difference = 0.01, 95% CI [-0.08 to 0.09], Standard Error of Mean 0.043
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; This statistical analysis is for pain/discomfort; Test type: Superiority or Other; p = 0.1628, ANCOVA; [statistical method as in outcome 7, analysis 1]; least squares mean difference = -0.06, 95% CI [-0.14 to 0.02], Standard Error of Mean 0.043
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; This statistical analysis is for anxiety/depression; Test type: Superiority or Other; p = 0.4654, ANCOVA; [statistical method as in outcome 7, analysis 1]; leaset squares mean difference = 0.03, 95% CI [-0.05 to 0.10], Standard Error of Mean 0.037
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; This statistical analysis is for Dolan 1997 Index score; Test type: Superiority or Other; p = 0.5000, ANCOVA; [statistical method as in outcome 7, analysis 1]; least squares mean difference = 0.01, 95% CI [-0.02 to 0.04], Standard Error of Mean 0.017
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; This statistical analysis is for Dolan 2001 Index Score; Test type: Superiority or Other; p = 0.5493, ANCOVA; [statistical method as in outcome 7, analysis 1]; leaset squares mean difference = -0.02, 95% CI [-0.07 to 0.04], Standard Error of Mean 0.026

8. Secondary Outcome: Baseline Scores in the Medical Outcomes Study Sleep Scale (MOS-SS) - Sub-domain Score.
Description: MOS-SS is a self administered measure consisting of twelve items that assess the key constructs of sleep. Instrument scored results in 7 subscales: sleep disturbance, snoring, awaken short of breath or with headache, quantity of sleep, optimal sleep, sleep adequacy, somnolence. Two index measures that assess sleep disturbance was also constructed to provide composite scores.
  Sleep disturbance, snoring, somnolence, awaken short of breath, and the 9 items sleep problems index all have score ranges from 0 (no sleep problems) to 100 (greater sleep problems), therefore a negative change indicates improvement.
  Sleep adequacy is scored 0 (least sleep adequacy) to 100 (better sleep adequacy), therefore a positive change indicates improvement.
  Quantity of sleep is scored 0 (less quantity of sleep) to 24 (greater quantity of sleep), therefore a positive change indicates improvement.
  Optimal sleep is scored Yes if average hours of sleep is in range of 7-8 hours.
Time Frame: Baseline
Population: ITT population: all randomized participants who took at least one dose of study drug.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Units on a scale
  Sleep Disturbance Score (N = 274, 265) | 42.50 (25.791) [0 to 100] | 43.75 (25.080) [0 to 100]
  Sleep Adequancy Score (N = 274, 265) | 40.0 (28.153) [0 to 100] | 40.0 (28.582) [0 to 100]
  Snoring Score (N = 272, 263) | 20.0 (33.482) [0 to 100] | 20.0 (34.084) [0 to 100]
  Awaken Short of Breath Score (N = 274, 265) | 0.0 (25.647) [0.0 to 100] | 0.0 (21.541) [0.0 to 100]
  Quantity of Sleep Score (hours) (N = 273, 265) | 6.0 (1.360) [2.0 to 10.0] | 6.0 (1.411) [2.0 to 10.0]
  Somnolence Score (N = 274, 265) | 26.67 (21.618) [0.0 to 100] | 26.67 (19.884) [0.0 to 100]
  Sleep Problem Index (9) Score (N = 274, 265) | 40.56 (20.282) [0.0 to 88.3] | 41.11 (19.720) [0.0 to 88.9]
  Optimal Sleep Score (N = 273, 265) | 0.0 (0.476) [0.0 to 1.0] | 0.0 (0.487) [0.0 to 1.0]

9. Secondary Outcome: Mean Change From Baseline in the Medical Outcomes Study Sleep Scale (MOS-SS) - Sub-domain Score.
Description: as for outcome 8
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Units on a scale
  Sleep Disturbance Score (N = 257, 245) | -14.71 [-17.57 to -11.85] | -11.24 [-14.16 to -8.33]
  Sleep Adequancy Score (N=257, 245) | 10.13 [6.49 to 13.76] | 8.16 [4.43 to 11.89]
  Snoring Score (N = 257, 245) | -2.22 [-5.46 to 1.03] | -3.27 [-6.59 to 0.04]
  Awaken Short of Breath Score (N = 257, 245) | -3.61 [-6.30 to -0.92] | -3.03 [-5.78 to -0.27]
  Quantity of Sleep Score (hours) (N = 257, 245) | 0.42 [0.19 to 0.66] | 0.26 [0.03 to 0.50]
  Somnolence Score (N = 257, 245) | -1.61 [-3.99 to 0.77] | -3.74 [-6.17 to -1.31]
  Sleep Problem Index (9) Score (N = 257, 245) | -9.86 [-12.17 to -7.56] | -8.19 [-10.55 to -5.83]
  Optimal Sleep Score (N = 256, 245) | 0.11 [0.05 to 0.18] | 0.04 [-0.03 to 0.10]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis for Sleep Disturbance Score; Test type: Superiority or Other; p = 0.0545, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = 3.5, 95% CI [-0.07 to 7.00], Standard Error of Mean 1.80
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis for Sleep Adequancy Score; Test type: Superiority or Other; p = 0.3913, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = -2.0, 95% CI [-6.47 to 2.54], Standard Error of Mean 2.29
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis for Snoring Score; Test type: Superiority or Other; p = 0.6059, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = -1.1, 95% CI [-5.06 to 2.96], Standard Error of Mean 2.04
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis for Awaken Short of Breath Score; Test type: Superiority or Other; p = 0.7317, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = 0.6, 95% CI [-2.76 to 3.93], Standard Error of Mean 1.70
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis for Quantity of Sleep Score (hours); Test type: Superiority or Other; p = 0.2663, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = -0.2, 95% CI [-0.45 to 0.12], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Pregabalin; Statistical analysis for Somnolence Score; Test type: Superiority or Other; p = 0.1562, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = -2.1, 95% CI [-5.08 to 0.82], Standard Error of Mean 1.50
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis for Sleep Problem Index (9) Score; Test type: Superiority or Other; p = 0.2490, ANCOVA; [statistical method as in outcome 7, analysis 1]; least square mean difference = 1.7, 95% CI [-1.18 to 4.53], Standard Error of Mean 1.45
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis for Optimal Sleep Score; Test type: Superiority or Other; p = 0.0609, ANCOVA; [statistical method as in outcome 7, analysis 1]; leaet squares mean difference = -0.1, 95% CI [-0.15 to 0.00], Standard Error of Mean 0.04

10. Secondary Outcome: Percentage of Participants in MOS-SS With Optimal Sleep Status.
Description: MOS-SS optimal sleep status analyzed on a scale of four parameters: any improvements, no change, any worsening and not applicable.
Time Frame: Week 15
Population: ITT population: all randomized subjects who took at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Percentage of participants
  Any Improvements | 21.2 | 18.5
  No Change | 66.1 | 60.8
  Any Worsening | 6.2 | 13.2
  Not applicable | 6.6 | 7.5
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.7165, Cochran-Mantel-Haenszel — p-values based on CMH test stratified by pooled center and trauma type, patients with unknown status at baseline or endpoint will not be included in the calculation of p-values

11. Secondary Outcome: Percentage of Responders to Treatment With Pregabalin Measured as Reduction in Mean Pain Score of ≥30%.
Description: Participants with at least 30% reduction in the mean pain score from baseline to each week. Weekly mean pain NRS scores are derived from the daily pain NRS and calculated as the mean of the available scores in the 7 days. Generally, week 'n' mean pain score is defined as the mean of the 7 daily diary pain ratings from Day 2+7*(n-1) to Day 1+7*n. At least 4 entries within the last 7 days are required to calculate a mean score. Scores range from 0 (no pain) to 10 (worst possible pain), with higher scored indicating increased pain.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Percentage of participants
  Week 1 (N = 260, 258) | 11.92 | 5.04
  Week 2 (N = 254, 244) | 27.17 | 20.08
  Week 3 (N = 252, 245) | 38.89 | 30.20
  Week 4 (N = 246, 229) | 41.87 | 34.50
  Week 5 (N = 241, 226) | 45.64 | 38.05
  Week 6 (N = 244, 227) | 48.77 | 41.41
  Week 7 (N = 240, 216) | 49.58 | 43.06
  Week 8 (N = 236, 213) | 50.42 | 46.48
  Week 9 (N = 232, 214) | 50.86 | 47.66
  Week 10 (N = 229, 212) | 52.84 | 47.17
  Week 11 (N = 231, 211) | 52.38 | 51.18
  Week 12 (N = 227, 209) | 54.63 | 52.63
  Week 13 (N = 226, 204) | 57.08 | 54.41
  Week 14 (N = 223, 208) | 57.40 | 54.33
  Week 15 (N = 196, 187) | 57.65 | 58.29
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 1; Test type: Superiority or Other; p = 0.0028, Gen linear model-logistic link function; Model terms include categorical: treatment, center, trauma type, week, and treatment-by-week interaction; and continuous: baselines mean pain score; Odds Ratio (OR) = 3.20, 95% CI [1.50 to 6.86]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 2; Test type: Superiority or Other; p = 0.0360, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI [1.03 to 2.68]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 3; Test type: Superiority or Other; p = 0.0235, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI [1.07 to 2.45]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 4; Test type: Superiority or Other; p = 0.0619, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI [0.98 to 2.24]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 5; Test type: Superiority or Other; p = 0.0677, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI [0.97 to 2.20]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0707, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI [0.97 to 2.16]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 7; Test type: Superiority or Other; p = 0.1313, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI [0.91 to 2.06]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 8; Test type: Superiority or Other; p = 0.3072, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI [0.82 to 1.86]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 9; Test type: Superiority or Other; p = 0.3947, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI [0.79 to 1.80]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 10; Test type: Superiority or Other; p = 0.1462, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI [0.90 to 2.05]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 11; Test type: Superiority or Other; p = 0.6854, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI [0.72 to 1.64]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.5025, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI [0.76 to 1.74]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 13; Test type: Superiority or Other; p = 0.4908, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI [0.76 to 1.76]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 14; Test type: Superiority or Other; p = 0.4245, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI [0.78 to 1.80]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 15; Test type: Superiority or Other; p = 0.8464, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI [0.61 to 1.49]

12. Secondary Outcome: Percentage of Responders to Treatment With Pregabalin Measured as Reduction in Mean Pain Score of ≥50%
Description: Participants with at least 50% reduction in the mean pain score from baseline to each week. Weekly mean pain NRS scores are derived from the daily pain NRS and calculated as the mean of the available scores in the 7 days. Generally, week 'n' mean pain score is defined as the mean of the 7 daily diary pain ratings from Day 2+7*(n-1) to Day 1+7*n. At least 4 entries within the last 7 days are required to calculate a mean score. Scores range from 0 (no pain) to 10 (worst possible pain), with higher scored indicating increased pain.
Time Frame: Week 15
Population: ITT population: all randomized participants who took at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 274 | 265
Percentage of participants
  Week 1 (N = 260, 258) | 4.62 | 2.33
  Week 2 (N = 254, 244) | 11.42 | 6.97
  Week 3 (N = 252, 245) | 22.62 | 13.47
  Week 4 (N = 246, 229) | 25.20 | 17.90
  Week 5 (N = 241, 226) | 28.22 | 19.47
  Week 6 (N = 244, 227) | 29.51 | 22.91
  Week 7 (N= 240, 216) | 30.42 | 22.22
  Week 8 (N = 236, 213) | 33.05 | 27.70
  Week 9 (N = 232, 214) | 34.05 | 26.17
  Week 10 (N = 229, 212) | 32.75 | 26.42
  Week 11 (N = 231, 211) | 34.20 | 25.59
  Week 12 (N = 227, 209) | 37.89 | 26.79
  Week 13 (N = 226, 204) | 35.84 | 27.45
  Week 14 (N = 223, 208) | 37.67 | 29.81
  Week 15 (N = 196, 187) | 39.80 | 34.22
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 1; Test type: Superiority or Other; p = 0.1633, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI [0.74 to 6.00]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 2; Test type: Superiority or Other; p = 0.0652, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI [0.96 to 3.85]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 3; Test type: Superiority or Other; p = 0.0039, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI [1.29 to 3.77]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 4; Test type: Superiority or Other; p = 0.0382, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI [1.03 to 2.83]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 5; Test type: Superiority or Other; p = 0.0137, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.86, 95% CI [1.14 to 3.05]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 6; Test type: Superiority or Other; p = 0.0693, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI [0.97 to 2.49]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 7; Test type: Superiority or Other; p = 0.0349, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI [1.04 to 2.73]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 8; Test type: Superiority or Other; p = 0.1227, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI [0.91 to 2.29]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 9; Test type: Superiority or Other; p = 0.0364, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI [1.03 to 2.63]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 10; Test type: Superiority or Other; p = 0.0667, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI [0.97 to 2.49]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 11; Test type: Superiority or Other; p = 0.0176, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI [1.10 to 2.84]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0030, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI [1.27 to 3.23]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 13; Test type: Superiority or Other; p = 0.0256, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI [1.07 to 2.74]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 14; Test type: Superiority or Other; p = 0.0314, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI [1.05 to 2.64]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 15; Test type: Superiority or Other; p = 0.1889, Gen linear model-logistic link function; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI [0.85 to 2.21]

ADVERSE EVENTS:
Time Frame: From Day -21 to Day 112 (week 16) i.e. from baseline until 1 day post last taper dose.
Description: The adverse events reporting period was from the signing of the informed consent (at screening) throughout the study including 28 calendar days from the last dose of study medication.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/274 | 7/265
Other Adverse Events (participants affected / at risk) | 75/274 | 33/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=274) | Placebo (N=265)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=274) | Placebo (N=265)
Nausea (Gastrointestinal disorders) | 14 (15) | 8 (8)
Fatigue (General disorders) | 14 (16) | 10 (10)
Dizziness (Nervous system disorders) | 40 (51) | 11 (13)
Somnolence (Nervous system disorders) | 27 (31) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.